CLINICAL TRIAL: NCT01559922
Title: A Phase 3 Randomized Placebo-Controlled Double-Blind Study of the Use of Artefill® for Moderate to Severe Atrophic Acne Scar Correction
Brief Title: Use of Artefill® for Moderate to Severe Atrophic Acne Scar Correction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suneva Medical, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUN-11-001
Record Dates: First submitted 2012-03-15; First posted 2012-03-21 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2016-12

CONDITIONS: Atrophic Acne Scar
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Normal Saline
- Artefill (Experimental): Dermal Filler
  Interventions: Device: Artefill

INTERVENTIONS:
Drug: Normal Saline — Administration of up to 2 study treatments administered 6 weeks apart
  Arms: Placebo
Device: Artefill — Administration of up to 2 study treatments administered 6 weeks apart
  Arms: Artefill

SUMMARY:
The purpose of this study is to determine whether Artefill is safe and effective for the correction of atrophic facial acne scars.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study assessing the efficacy and safety of Artefill for correction of moderate to severe atrophic acne scars.

The study is divided into two study periods. In Period I, scars meeting the treatment criteria will be individually identified, numbered and mapped using photographs and transparent sheets prior to treatment. This mapping will be used to track individual scars throughout the trial. Four (4) weeks following a baseline qualification visit, subjects randomized to treatment will receive one treatment of Artefill or Control (saline), administered by the Treating Investigator. At 72 hours following injections, subjects will be followed-up by telephone to confirm the occurrence of any AEs. Subjects will return to the clinic at 2 weeks for follow-up evaluation, and then at 4 weeks where subjects may receive one optional touch-up treatment. Subjects receiving touch-up treatment will be followed-up by telephone at 72 hours to confirm the occurrence of any AEs, and return for clinic visits at 6 weeks and 8 weeks. All subjects will then return for clinic follow-up at months 3 and 6 (after last treatment).

Period II is open label and will begin at month 6. Artefill group subjects will return to the clinic for assessments at months 9 and 12 (Track A) and Control group subjects will enter Track B, re-establish baseline, and complete additional month 6 visit activities including Artefill treatment. Subjects will receive touch up (if required) 4 weeks later, and be followed for an additional 12 months.

Subjects will be required to abstain from other aesthetic treatment to their face during the study period and failure to do so will be considered a protocol violation. However, if a subject does receive additional aesthetic or non-aesthetic treatments, available information on such treatment will be collected and the subject will be continued to be followed per protocol. Such subjects will not be excluded from the analysis, but will also be evaluated separately.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be an outpatient, male or female subjects of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study.
2. Subject must have moderate to severe atrophic acne scars
3. Subject must desire correction of his/her moderate to severe acne scarring.
4. Subjects of all Fitzpatrick skin types are eligible.
5. Subject must be willing to withhold additional aesthetic therapies to the face (eg, other soft tissue fillers: Restylane, Radiesse, Sculptra, and/or any resurfacing procedures for the duration of the study.
6. Subject must be able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
7. Subject must sign an IRB-approved Informed Consent form, Photographic Release Form, and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed

Exclusion Criteria:

1. Female subjects that are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
2. Undergo facial treatments with any listed of the prohibited treatment/procedures and/or use of any other prohibited treatment/procedure within certain time periods.
3. Have any skin pathology or condition that could interfere with the evaluation of the treatment areas, worsen due to the proposed treatment or require interfering topical, systemic or surgical therapy.
4. Have a recent or current history of inflammatory skin disease, infection, cancerous/pre-cancerous lesion, unhealed wound or clinically significant acne in the proposed treatment areas. Clinically significant acne is defined as a patient whom has >3 active inflammatory acne lesions in either the right or left treatment area.
5. Have a history of systemic granulomatous diseases active or inactive (eg, Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (eg, lupus, dermatomyositis, etc.).
6. Have hypertrophic acne scars, any evidence of keloid scarring, predominantly icepick scarring (defined as more than half of all scar area in either the left or right or treatment area) or sinus tract scars.
7. Have a known hypersensitivity or previous allergic reaction to any of the components of the study device (including lidocaine or any amide-based anesthetic), or has a history of allergies to any bovine collagen products, including but not limited to injectable collagen, collagen implants, hemostatic sponges, and collagen-based sutures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Serreta, Study Director — Suneva Medical
Locations (10):
- United States (10):
  - Call Suneva for Info, Beverly Hills, California
  - Call Suneva for Info, Los Angeles, California
  - Call Suneva for Info, San Diego, California
  - Call Suneva for Info, Santa Monica, California
  - Call Suneva for Info, Miami Beach, Florida
  - Call Suneva for Info, St. Petersburg, Florida
  - Call Suneva for Info, Glenn Dale, Maryland
  - Call Suneva for Info, Wellesley, Massachusetts
  - Call Suneva for Info, Houston, Texas
  - Call Suneva for Info, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 199 subjects were enrolled into the Screening phase. 175 subjects were randomized, with a total of 147 subjects receiving study treatment. Data presented are from all Randomized/Treated subjects (i.e., n=147).
Period: Overall Study
Arm/Group | Placebo | Artefill
Started | 50 | 97
Completed | 46 | 87
Not Completed | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Artefill | Total
Number analyzed (Participants) | 50 | 97 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 97 | 147
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 60 | 90
  Male | 20 | 37 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 20 | 28
  White | 38 | 70 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 20 | 33
  Not Hispanic or Latino | 37 | 77 | 114
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 97 | 147

OUTCOME MEASURES:

1. Primary Outcome: ASRS Responder Rate at 6 Months
Description: Subject considered to be a "responder" if at least 50% of treated scars demonstrate an ASRS improvement of ≥ 2-point (Blinded Evaluator assessment).
Time Frame: 6 months post-treatment
Population: Full Analysis Population included only subjects that passed screening
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Artefill
Number analyzed (Participants) | 50 | 97
percentage of participants | 32.4 [17.3 to 52.2] | 67.4 [51.3 to 80.2]

ADVERSE EVENTS:
Time Frame: 12 months post treatment
Arm/Group | Placebo | Artefill
Serious Adverse Events (participants affected / at risk) | 2/50 | 3/97
Other Adverse Events (participants affected / at risk) | 0/50 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Artefill (N=97)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast Cancer (recurrent) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Suneva, as the Sponsor, has a proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation among multiple investigators and sites and Suneva personnel. Authorship will be established prior to the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multi-center study except as agreed with Suneva.